CLINICAL TRIAL: NCT04968444
Title: The Bespoke One-Off Spinal Treatment (BOOST) Workshop Versus Traditional 1:1 Physiotherapy Care for the Management of Hospital Staff With Chronic Spinal Pain: A Randomised Controlled Trial
Brief Title: BOOST Workshop Versus Traditional 1-1 Physiotherapy for Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 247300
Record Dates: First submitted 2020-12-03; First posted 2021-07-20 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-05

CONDITIONS: Back Pain
Keywords: occupational health; physiotherapy; sickness
MeSH Terms: conditions — Back Pain | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: blinding of investigator through masking of participant identified to each group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- one to one traditional physiotherapy (Active Comparator): For clarity, 1-1 physiotherapy takes the form of a private consultation between patient and therapist. A discussion of symptoms is had and an individual physical examination is undertaken to explore what is mechanically causing their pain and what can be offered to help. This is also when the initial outcome scores are taken. Treatments are then offered which can take the form of exercise therapy, massage, and manual therapy. Symptoms are regularly monitored for effectiveness of treatment and adjusted accordingly. The number of sessions that forms their treatment is variable depending on response to treatment and how they are coping. At the final session the end outcome scores will be taken.
  Interventions: Other: Physiotherapy
- BOOST workshop group (Active Comparator): The BOOST workshop is a novel approach whereby participants are invited to a 2.5 hour interactive session. Subjective discussion at the start is had about how people are affected and impacted by their back pain, and outcome scores are completed. Then during the 2.5 hours there is a delivery of information and a practical exercise component to better inform the participants on how to manage their back pain and understand it better. Following this on 3 separate occasions, 1 month apart further top up information is sent to ensure they remember exercises and advice on practical management if a flare up occurs or they are struggling to fit activity in to day to day routines. Finally, at 3 months, there participants are invited back to complete the outcomes scores but also to discuss any concerns they are having and be given any advice to support them continuing with managing with any ongoing symptoms.
  Interventions: Other: Back Pain Workshop

INTERVENTIONS:
Other: Physiotherapy — Physiotherapy helps to restore movement and function when someone is affected by injury, illness or disability. It can also help to reduce your risk of injury or illness in the future.
  This can take the form of
  * advice and education
  * manual therapy
  * exercise prescription
  * relaxation
  Arms: one to one traditional physiotherapy
Other: Back Pain Workshop — Back workshop is an intervention protocol consisting of an educational program and skills acquisition program, including physical exercises. The session is supervised by a specialist physiotherapist.
  Arms: BOOST workshop group

SUMMARY:
This research is aiming to address whether a group workshop is a more superior treatment to traditional physiotherapy for the management of back pain in a hospital workforce. In the UK during 2016-17, 31.2 million work days were lost due to work-related ill health and injury. Of these 8.9 million were down to musculoskeletal disorders. This equated to 17.6 days per person. In the general population, the reports of low back pain have been as high as 36% of adults with a first occurrence. In an adult's lifetime, the prevalence of chronic low back pain is about 23%. This makes the importance of managing these conditions of great importance. And the impact to a working population is great, in respects to work satisfaction, sickness and absenteeism. Significance should also be placed on the impact this has to the individual, with regards to their health and wellbeing.

The participants will be taken from NHS staff working within the hospital environment and that self-refer internally for physiotherapy into the Trust's Occupational Health Service. Once the participants are accepted in Occupational Health Physiotherapy, they are managed as staff requiring physiotherapy and not at 'patients'. There is no contact with their primary care practitioner. For the study, participants will either receive traditional one to one physiotherapy or a bespoke one off workshop. All of the participants will be followed up 3 months after their treatment has finished.

DETAILED DESCRIPTION:
Traditionally, treatment for chronic pain, and back pain in particular has been on exercise and education. Back schools and multi-speciality classes are evidence based effective management recommended to this population (Heymans et al, 2004; Airaksinen et al, 2006). However, for a busy NHS Trust, staff taking time out of their week for 6-12 weeks would not be practical or supportive to patient care and work-life balance. Therefore a one-off seminar based lecture and interactive workshop would be using less clinical time for the staff to attend and may be better for both the individual and the organisation.

The importance of piloting a novel method of delivering treatment to this cohort is to ensure that the content is supported by the current evidence. A Cochrane review (Cochrane 2004) found moderate evidence that Back Schools in an occupational setting can reduce pain and increase functional and return to work status in the short and intermediate term. Waddal's review (2001) also supports this idea, stating the some form of back school or MDT (multidisciplinary team) rehabilitation at the sub-acute stage has produced faster recovery. The Kamper study (2015) concluded that MDT delivery of care was better than physical treatment in the occupational setting for back pain management. There is therefore no clear affirmative support for a specific method of care delivery but having a group environment of similar pathology and using an MDT skill mix is recommended.

The Occupational Health Model of care within this setting is aiming to deliver bespoke information to specific cohorts of staff and pathologies with the long term aim of self-management and injury prevention. Waddel et al (2004) has suggested innovative education approaches for prevention and management, specifically designed to overcome psycho-social issues and encourage responsibility for their own care. Therefore a successful intervention should encapsulate these ideas.

As there is little research into the novel approach of delivering seminar-style MDT education and advice to a cohort of staff, this pilot will assess the effect of this intervention.

The purpose of this research is to compare the effectiveness of 2 interventions for the management of chronic spinal pain in staff members based in a hospital setting. The primary aim is to establish the most effective method of management for this sub group of staff. This research came from service user feedback and management issues around staff having to take considerable amount of time away from clinical activity. And the trend noticed in the Trust for increasing back pain referrals. Therefore, the investigators were looking at a way that could make an intervention effective and have minimal impact on staff being away from their work duties. However, the results of this study will inform practice for the best management for back pain across all working populations and therefore can be generalizable outside of this selected target group.

For recruitment to the study, The Occupational Health Physiotherapy service is routinely advertised on the Trust intranet webpage (internal staff site) and at roadshows and Trust induction. The research team would not be advertising our study but making staff aware when the referral is received that the team are running and trial and that they have been allocated to attend one of the two group.

When the staff member is contacted by phone and booked into their session, the participant will be emailed confirmation of the appointment details and the participant information sheet. Each participant will be advised that they can change their mind about treatment allocation up to the day of appointment and tehe investigator would be gaining signed consent at this time so they have up to 2 weeks to decide. Witnessed consent will be gained at the initial meeting either in the workshop or in the initial one to one session. All staff at GSTFT speak English and therefore should be able to independently read and sign any information and forms.

The inclusion/exclusion criteria are as follows:

Inclusion criteria:

1. Staff member of GSTFT
2. New referral with a history of spinal pain (cervical/ thoracic/ lumbar) for more than 3 months
3. Consents to attend 2 sessions - seminar and follow up if in BOOST workshop, or complies with one to one treatment as outlined by the treating therapist.

Exclusion criteria:

1. Acute spinal pain - that of 6 weeks or less
2. Had treatment for the condition of chronic spinal pain in last 6 months as may still be gaining treatment benefits from this and unclear if change was due to our interventions

This project has been discussed at Occupational Health roadshows run in the Trust and staff have been asked for feedback on the plans for the project. All are in favour of a multi-disciplinary approach and the contact with staff is favourable. There was concern about the meaning of 'traditional physiotherapy'. This was explained that all those in this group would have a tailored treatment programme dependent on assessment. Staff were also concerned about being allowed to attend appointments and the possibility that they may have to miss some. The investigators explained that there is no requirement for compliance due to the nature of the intervention - the BOOST workshop is a one-off intervention and the 1-1 treatment group is routine physiotherapy care. All non-attendance will be noted and reported in the project analysis.

The data to be collected will be as follows:

Pre-intervention - all at baseline

* Patient demographics - age, sex, work-type classification (from patient referral form)
* Sickness absence (in last 3 months) (from initial data collection questionnaire)
* Numerical rating scale for pain (NRS) (from initial data collection questionnaire)
* Patient specific functional scale (PSFS) (from initial data collection questionnaire)
* Patient-activation measure (from initial data collection questionnaire)
* StarT Back (screening tool for sub-group analysis). (from initial data collection questionnaire)

Post-intervention

* Sickness absence (in last 3 months) (from final contact/follow up data collection questionnaire)
* Numerical rating scale for pain (from final contact/follow up data collection questionnaire)
* Patient specific functional scale (from final contact/follow up data collection questionnaire)
* Service evaluation questionnaire (from final contact/follow up data collection questionnaire)
* Patient-activation measure (from final contact/follow up data collection questionnaire)

The treating/intervention therapist will issue the questionnaire/data collection sheet for the participant to complete. This is then handed to the administrative staff for entry on the central database to support reducing risk of bias.

Sickness absence, NRS and PSFS are all validated outcomes to show change over time and occupational improvement following an intervention. StarT Back is a stratification tool only taken at initial contact to sub-group the participant in relation to their back pain. This is for us to analyse the most likely group to respond to each intervention as a possible variable to outcome.

ELIGIBILITY:
The inclusion/exclusion criteria are as follows:

Inclusion criteria:

1. Staff member of GSTFT
2. New referral with a history of spinal pain (cervical/ thoracic/ lumbar) for more than 3 months
3. Consents to attend 2 sessions - seminar and follow up if in BOOST workshop, or complies with one to one treatment as outlined by the treating therapist.

Exclusion criteria:

1. Acute spinal pain - that of 6 weeks or less
2. Had treatment for the condition of chronic spinal pain in last 6 months as may still be gaining treatment benefits from this and unclear if change was due to our interventions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2023-04-01 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
The Keele STarT Back Screening tool | Baseline
  score out of 9, for low, medium of high risk of chronicity of back pain

SECONDARY OUTCOMES:
Numerical rating score | baseline and at 3 months following this
  scale 0-10 rating pain levels, 0 no pain and 10 worst pain
Patient Specific Functional Score | baseline and at 3 months following this
  Rate of difficulty in managing certain tasks rated at 0-10, 0 full disability and 10 no problems
sickness | baseline and at 3 months following this
  number of days sick in last 90 days

IPD SHARING:
Plan to Share IPD: No
This is an individual study on a single site. No plan to share as information is confidential